CLINICAL TRIAL: NCT04501276
Title: A Phase 1b/2, Open-Label, Dose Escalation and Expansion Study of ADG116, ADG116 Combined With Toripalimab (Anti-PD-1 Antibody), ADG116 Combined With ADG106 (Anti-CD137 Antibody) in Patients With Advanced/Metastatic Solid Tumors
Brief Title: A Phase 1b/2 Study of ADG116, ADG116 Combined With Anti-PD-1 Antibody or Anti-CD137 Antibody in Solid Tumors Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adagene Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADG116-1003
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Advanced/Metastatic Solid Tumors
Keywords: Advanced/Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A : Dose escalation of ADG116 monotherapy (Experimental)
  Interventions: Drug: ADG116
- Part B : Dose escalation of ADG116 combined with anti PD1 drug (Experimental)
  Interventions: Drug: ADG116; Drug: anti PD1 drug
- Part C : Dose escalation of ADG116 combined with ADG106 (Experimental)
  Interventions: Drug: ADG116; Drug: ADG106

INTERVENTIONS:
Drug: ADG116 — For monotherapy ADG116 (Part A), ADG116 will be administered IV over 60 90 minutes until disease progression, intolerable toxicities, or withdrawal of consent, or up to 2 years.
Drug: ADG106 — For the ADG116-ADG106 combination regimen, ADG116 and ADG106 will be administered until disease progression, intolerable toxicities, or withdrawal of consent, or up to 2 years.
  Arms: Part C : Dose escalation of ADG116 combined with ADG106
Drug: anti PD1 drug — For the ADG116-anti PD1 combination regimen, ADG116 and anti PD1 will be administered until disease progression, intolerable toxicities, or withdrawal of consent, or up to 2 years.
  Arms: Part B : Dose escalation of ADG116 combined with anti PD1 drug

SUMMARY:
This is a Phase 1, open-label, dose escalation study in patients with advanced/metastatic solid tumors. Study drug, ADG116, is an anti -CTLA-4 fully human monoclonal antibody that specifically binds to human CTLA-4. ADG106, a fully human ligand-blocking agonistic anti-CD137 IgG4 mAb, is expected to enhance the activity of activated T cells. The enhanced antitumor efficacy results observed from the preclinical studies of ADG116 in combination with ADG106 or anti-PD-1 provided further support to explore such combinations in clinical settings for better patient responses.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

1. ≥ 18 years of age at the time of informed consent.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
3. Patients with advanced or metastatic solid tumors, who have progressed after all standard therapies, or for whom no further standard therapy exists.
4. At least 1 measurable lesion at baseline according to the definition of RECIST v1.1.
5. Adequate organ function.

Exclusion Criteria:

• Patients who meet any of the following criteria cannot be enrolled:

1. Pregnant or breastfeeding females.
2. Childbearing potential who does not agree to the use of contraception during the treatment period..
3. Treatment with any investigational drug within washout period.
4. Grade ≥ 3 immune-related AEs (irAEs) or irAE that lead to discontinuation of prior immunotherapy.
5. Central nervous system disease involvement
6. History or risk of autoimmune disease.
7. History of life-threatening hypersensitivity or known to be allergic to protein drugs or recombinant proteins or any ingredients contained in the ADG116 drug formulation.
8. Patients requiring systemic treatment with corticosteroids
9. Patients receiving granulocyte colony stimulating factor (G-CSF), within 14 days prior to the first dose of the study drug.
10. Any uncontrolled active infections requiring systemic antimicrobial treatment (viral, bacterial, or other), or uncontrolled or poorly controlled, asthma, chronic obstructive pulmonary disease (COPD).
11. Major surgery within 4 weeks prior to the first dose of the study drug.
12. Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing dose-limiting toxicities escalating dose levels in adults with advanced / metastatic solid tumors | From first dose of ADG116 (Week 1 Day 1) until 21 days
Number of participants with adverse events as assessed by CTCAE v5.0 | From first dose of ADG116 (Week 1 Day 1) to 28 days post last dose

SECONDARY OUTCOMES:
Area under the time concentration curve (AUC) from time zero to infinity (AUC0-inf) | From first dose (Cycle 1 Day 1, ) until the last dose (up to 2 years)
Maximum (peak) plasma concentration (Cmax) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
Time to maximum (peak) plasma concentration (Tmax) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
Trough plasma concentration (Ctrough) | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
Incidence of ADAs | From first dose (Cycle 1 Day 1,) until the last dose (up to 2 years)
Preliminary evidence of antitumor activity as characterized by objective response rate (ORR), disease control rate (DCR), duration of response (DOR), duration of stable disease, progression free survival (PFS), and overall survival (OS). | From first dose of ADG116 (Week 1 Day 1) to 28 days post last dose

CONTACTS AND LOCATIONS:
Locations (4):
- Next Oncology, San Antonio, Texas, United States
- Australia (3):
  - Ashford Cancer Centre Research, Kurralta Park
  - Cabrini Hospital, Malvern
  - Macquarie University, Sydney

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brahmer JR, Lacchetti C, Schneider BJ, Atkins MB, Brassil KJ, Caterino JM, Chau I, Ernstoff MS, Gardner JM, Ginex P, Hallmeyer S, Holter Chakrabarty J, Leighl NB, Mammen JS, McDermott DF, Naing A, Nastoupil LJ, Phillips T, Porter LD, Puzanov I, Reichner CA, Santomasso BD, Seigel C, Spira A, Suarez-Almazor ME, Wang Y, Weber JS, Wolchok JD, Thompson JA; National Comprehensive Cancer Network. Management of Immune-Related Adverse Events in Patients Treated With Immune Checkpoint Inhibitor Therapy: American Society of Clinical Oncology Clinical Practice Guideline. J Clin Oncol. 2018 Jun 10;36(17):1714-1768. doi: 10.1200/JCO.2017.77.6385. Epub 2018 Feb 14. PMID 29442540
- [Background] Melero I, Hervas-Stubbs S, Glennie M, Pardoll DM, Chen L. Immunostimulatory monoclonal antibodies for cancer therapy. Nat Rev Cancer. 2007 Feb;7(2):95-106. doi: 10.1038/nrc2051. PMID 17251916
- [Background] Finn OJ. Immuno-oncology: understanding the function and dysfunction of the immune system in cancer. Ann Oncol. 2012 Sep;23 Suppl 8(Suppl 8):viii6-9. doi: 10.1093/annonc/mds256. PMID 22918931